CLINICAL TRIAL: NCT00040313
Title: A Phase II Randomized, Controlled, Double-Masked, Dose-Finding, Multi-Center, Comparative Trial, in Parallel Groups, to Establish the Safety and Preliminary Efficacy of Intravitreal Injections of EYE001 (Anti-VEGF Pegylated Aptamer), Given Every 6 Weeks for 12 to 30 Weeks to Patients With Clinically Significant Diabetic Macular Edema (CSME) Involving the Center of the Macula
Brief Title: Pegaptanib Sodium Compared to Sham Injection in Patients With DME Involving the Center of the Macula
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOP1005
Record Dates: First submitted 2002-06-24; First posted 2002-06-25 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — pegaptanib

INTERVENTIONS:
Drug: pegaptanib sodium (Macugen)

SUMMARY:
The purpose of the study is to determine whether pegaptanib sodium (Macugen) is safe and effective in slowing the leakage of fluid within the retina and thereby stabilizing or improving vision when compared to placebo injections. A total of 176 patients will be enrolled

ELIGIBILITY:
Inclusion Criteria:

Patients with clinically significant DME, VA 20/50-20/320 in the study eye and 20/100 in the fellow eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 2002-10; Study Completion 2005-02